CLINICAL TRIAL: NCT07118774
Title: The Effect of the Young Ambassadors Supporting Caregivers (YASC) Program: A Dual Randomized Controlled Trial
Brief Title: The Young Ambassadors Supporting Caregivers Program
Acronym: YASC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qi Wang, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SS5/31; SS5/31 (Other Grant/Funding Number: The University of Hong Kong)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Psychological Well-being; Caregiver Burden of Caregivers
Keywords: volunteer
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of this trial, neither the staff, university students and caregivers can be masked to allocation. The investigator data analyst will be blinded after study completion by having the intervention group information coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention: Mindfulness and Compassion Training (Experimental): Students randomly assigned to this group will receive 12 hours over 6 weeks (2-hour weekly sessions) teaching mindfulness meditation (e.g., loving-kindness, body scan) and compassion practices (e.g., self-compassion exercises). Content culturally adapted with Buddhist-influenced terminology and practices resonant with Hong Kong's context. Caregivers assigned to this group will receive students' help based on the mindfulness training.
  Interventions: Behavioral: Behavioral: mindfulness and compassion training
- Intervention: Caregiving Skills Training (Experimental): Students randomly assigned to this group will receive 12 hours over 6 weeks (2-hour weekly sessions) teaching including: Occupational therapist training (e.g., daily living support), Physical therapist training (e.g., safe transfers), Speech Therapist training (e.g., communication aids), and Registered Nurse training (e.g., vital signs monitoring), tailored to caregivers' needs. Caregivers assigned to this group will receive students' help based on the caregiver skills training.
  Interventions: Behavioral: Behavioral: caregiver skills training
- Control: Communication Skills Training (Active Comparator): Students randomly assiged to this group will receive 12 hours over 6 weeks (2-hour weekly sessions) focusing on active listening, empathy, and basic conversational skills, without specific mindfulness or caregiving techniques. Caregivers assigned to this group will receive students' help based on the communication skills training.
  Interventions: Behavioral: Behavioral: Communication skills training

INTERVENTIONS:
Behavioral: Behavioral: mindfulness and compassion training — Parallel randomized controlled trial
  Arms: Intervention: Mindfulness and Compassion Training
Behavioral: Behavioral: caregiver skills training — Parallel randomized controlled trial
  Arms: Intervention: Caregiving Skills Training
Behavioral: Behavioral: Communication skills training — Parallel randomized controlled trial
  Arms: Control: Communication Skills Training

SUMMARY:
This RCT will provide preliminary evidence on effective training for young adult volunteers to support older adult caregivers, addressing Hong Kong's aging crisis and caregiver burden. The objectives of this study include:

1. To examine the feasibility and acceptability of the interventions in Hong Kong's cultural context.
2. To evaluate the effects of three trainings (mindfulness/compassion, caregiving skills, communication skills) on young adult volunteers' preparedness for caregiving, meaning of life, and civic engagement.
3. To assess the impact of volunteer services on caregivers' depression, anxiety, and caregiver burden.

DETAILED DESCRIPTION:
This study will train 60 university students to provide volunteer services to 60 paired caregivers. The 60 university students will be assiged to receive three types of training as intervention arms:

* Intervention 1: Mindfulness and Compassion Training (n=20)

  o Training: 12 hours over 6 weeks (2-hour weekly sessions) teaching mindfulness meditation (e.g., loving-kindness, body scan) and compassion practices (e.g., self-compassion exercises). Content culturally adapted with Buddhist-influenced terminology and practices resonant with Hong Kong's context.
* Intervention 2: Caregiving Skills Training (n=20)

  o Training: 12 hours over 6 weeks (2-hour weekly sessions) teaching OT (e.g., daily living support), PT (e.g., safe transfers), ST (e.g., communication aids), and RN (e.g., vital signs monitoring) skills, tailored to caregivers' needs.
* Control: Communication Skills Training (n=20) o Training: 12 hours over 6 weeks (2-hour weekly sessions) focusing on active listening, empathy, and basic conversational skills, without specific mindfulness or caregiving techniques.

After the training, the students will be paired with 60 caregivers of older adults to apply what they have learned during the training to offer services to reduce the psychological burden of the caregivers.

ELIGIBILITY:
Volunteer Recruitment and Eligibility

This study will recruit university students in Hong Kong as youth volunteers. Eligible participants must meet the following criteria:

1. Aged 18-35 years;
2. Willing to complete training and commit to at least 2 hours of volunteer service per week for 6 weeks;
3. No self-reported major physical or mental health conditions, including cognitive impairment;
4. Limited prior formal volunteering experience (≤4 engagements in the past year).

Older Adult Caregiver Recruitment and Eligibility

We will recruit community-dwelling Chinese adults in Hong Kong who provide care for older adults. Eligible caregivers must:

1. Be aged 50 years or older;
2. Consent to interact with youth volunteers at least four times during the intervention;
3. Report no major physical or mental health conditions, including cognitive impairment; and
4. Have resided with and provided care for an older adult (aged 65+) for a minimum of one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Preparedness for Caregiving Scale | Baseline (pre-test), immediately post-test
  Preparedness for Caregiving Scale will be adopted to evaluate university student volunteers' self-perceived readiness to provide care across eight critical domains, including physical/emotional caregiving (e.g., "How well prepared are you to care for emotional needs?"), stress management, and emergency response. Each item is rated on a 5-point Likert scale (0=Not at all prepared to 4=Very well prepared), providing a quantitative measure of skill development through the intervention. Higher score indicate higher level of preparedness for caregiving skills. Total score ranged from 0 to 32.
Patient Health Questionnaire | Baseline (pre-test), immediately post-test
  This scale will be applied to caregivers of older adults who joined this study. The Patient Health Questionnaire (PHQ) is a widely used, self-administered screening instrument designed to facilitate the identification and assessment of common mental health disorders in clinical and research settings. Developed as part of the Primary Care Evaluation of Mental Disorders (PRIME-MD) project, the PHQ consists of several modules, each corresponding to specific psychiatric diagnoses according to DSM criteria. The most commonly used version, the PHQ-9, consists of nine items that assess the frequency of depressive symptoms over the past two weeks. Each item is scored on a four-point Likert scale (ranging from 0 = "not at all" to 3 = "nearly every day"), resulting in a total score ranging from 0 to 27. Higher scores indicate greater severity of depressive symptoms. The PHQ has demonstrated strong reliability and validity across diverse populations and is valued for its brevity, ease of use, an

SECONDARY OUTCOMES:
Civic Engagement Scale | Baseline (pre-test), immediately post-test
  This civic engagement scale will be adopted among volunteers to measure broader psychosocial outcomes through 14 items assessing attitudes (e.g., belief in community contribution) and behaviors (e.g., community participation frequency) on a 7-point scale (from 1 very disagee to 7 very agree). The score ranged from 14 to 98 with higher score indicate higher level of civic engagement. This scale demonstrated high reliability (α=0.80- 0.91) and validity in youth populations.
Meaning in Life Scale | Baseline (pre-test), immediately post-test
  Meaning in Life Scale will be adopted to assess volunteer' sense of purpose and fulfillment. This validated measure captures two key dimensions: the presence of meaning (e.g., "I understand my life's meaning") and the search for meaning (e.g., "I am seeking a deeper purpose in life"), rated on a Likert scale (typically 1=Strongly disagree to 7=Strongly agree). Total score ranged from 10 to 70 with higher score indicate higher level of meaning in life. Developed by Steger et al. (2006), the scale has demonstrated strong reliability (α=0.80+ for both subscales) and has been widely used in cross-cultural populations, including youth and older adults.
Generalized Anxiety Disorder scale | Baseline (pre-test), immediately post-test
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a brief, self-administered screening tool designed to assess the severity of generalized anxiety disorder symptoms over the previous two weeks. Developed by Spitzer et al. (2006), the GAD-7 consists of seven items, each rated on a four-point Likert scale ranging from 0 ("not at all") to 3 ("nearly every day"), resulting in a total score that ranges from 0 to 21. Higher scores indicate greater symptom severity. The GAD-7 has demonstrated strong reliability and validity in both clinical and general populations, and is widely used in research and primary care settings for screening, diagnosis, and monitoring of anxiety disorders.
Zarit Burden Interview | Baseline (pre-test), immediately post-test
  The Zarit Burden Interview 12-item version (ZBI-12) is a brief, self-administered questionnaire designed to assess the perceived burden of caregivers for individuals with chronic illnesses or disabilities. Adapted from the original 22-item ZBI, the ZBI-12 retains key items that capture multiple dimensions of caregiver strain, including emotional, social, and physical burden. Each item is rated on a 5-point Likert scale ranging from 0 ("never") to 4 ("nearly always"), resulting in a total score between 0 and 48, with higher scores indicating greater caregiver burden. The ZBI-12 has demonstrated good reliability and validity across diverse populations and is widely used in both research and clinical settings for the efficient assessment of caregiver stress.